CLINICAL TRIAL: NCT04272892
Title: An Investigation Into the Efficacy of Online Cognitive Behavioural Therapy for Insomnia ("Sleepio") to Improve Sleep After Stroke.
Brief Title: Improving Sleep in Rehabilitation After Stroke
Acronym: INSPIRES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Big Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INSPIRES
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2021-07

CONDITIONS: Stroke
Keywords: Sleep; Rehabilitation; Digital; Cognitive Behavioural Therapy for Insomnia
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants will be randomised (1:1 ratio) to the intervention or control group, using a computer generated minimisation method, with minimisation of between groups differences in age and baseline self-reported sleep quality (sleep condition indicator score)
Who Masked: Participant
Masking Description: Participants will be told that they will be assigned to one of two groups but will not be told whether one is hypothesised to be superior over another
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital CBT-I (Experimental): 6 weeks digital (online) cognitive behavioural therapy for insomnia
  Interventions: Behavioral: Digital cognitive behavioural therapy for insomnia
- Sleep hygiene information (Active Comparator): Leaflet of sleep hygiene information
  Interventions: Behavioral: Sleep hygiene information

INTERVENTIONS:
Behavioral: Digital cognitive behavioural therapy for insomnia — 6 weeks of cognitive behavioural therapy for insomnia (Sleepio) delivered online
  Other Names: Sleepio
  Arms: Digital CBT-I
Behavioral: Sleep hygiene information — A leaflet detailing advice to improve sleep through changes in sleep hygiene
  Arms: Sleep hygiene information

SUMMARY:
This study evaluates the efficacy of digital cognitive behavioural therapy for insomnia (Sleepio) in chronic stroke survivors. Half of the participants will receive access to the digital (online) programme, half will receive a leaflet with sleep hygiene information. The primary outcome will be changes in sleep quality, assessed as the score on the Sleep Condition Indicator.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of adult disability. Many stroke survivors report difficulties with sleep and our current research confirms this, indicating that chronic community dwelling stroke survivors experience poorer self-reported and objective sleep quality than age matched healthy controls.

"Sleepio" is an online Cognitive Behavioural Therapy for Insomnia (CBT-I) programme. The efficacy of this intervention has been demonstrated in people with chronic insomnia but has not yet been tested in people with stroke. The study therefore aims to determine whether digital CBT-I is effective for improving sleep quality in chronic stroke survivors. Participants will be randomised to receive either digital (online) CBT-I or a leaflet with sleep hygiene information. The primary outcome is the change in self-reported sleep quality, assessed using the Sleep Condition Indicator. Secondary outcomes include changes in sleep fragmentation and wake after sleep onset assessed with actigraphy, self-reported sleep onset latency from the sleep diaries, anxiety and depression using the PHQ9 and GAD7, quality of life using the SIS-8 and EQ-5D-5L as well as changes in healthcare costs during the 8 week follow up.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* At least 18 years of age
* At least 3 months post stroke
* Interest in improving sleep
* Can understand verbal and written English well enough to engage with the programme and study procedures (with assistance from carer if needed).
* Reliable access to internet
* Currently living in the United Kingdom
* Current stable health

Exclusion Criteria:

* Serious physical health concerns with surgery scheduled in the next 5 months
* Undergoing a psychological treatment programme for insomnia (with a health professional or online)
* Pregnancy
* Uncontrolled seizures
* Untreated diagnosed obstructive sleep apnoea
* Habitual night shift, evening or rotating shift-workers
* Other serious clinical condition that may affect participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Johansen-Berg, PhD, Principal Investigator — University of Oxford, UK
Locations (1):
- Wellcome Centre for Integrative Neuroimaging (WIN), Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified data are available upon reasonable request
Supporting Information: Study Protocol
Time Frame: Following publication of results
Access Criteria: Available upon reasonable request

REFERENCES:
- [Derived] Fleming MK, Smejka T, Macey E, Luengo-Fernandez R, Henry AL, Robinson B, Kyle SD, Espie CA, Johansen-Berg H. Improving sleep after stroke: A randomised controlled trial of digital cognitive behavioural therapy for insomnia. J Sleep Res. 2024 Apr;33(2):e13971. doi: 10.1111/jsr.13971. Epub 2023 Jul 5. PMID 37407096

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants failed to undergo the baseline assessment following consent, and were not randomised to group. Therefore, although 86 participants consented, the total started in the study when divided by group is 84
Period: Overall Study
Arm/Group | Digital CBT-I | Sleep Hygiene Information
Started | 48 | 36
Post-intervention Assessment | 35 | 33
Completed (8 week follow-up, defined as 8-weeks following the post-intervention assessment) | 34 | 33
Not Completed | 14 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Digital CBT-I | Sleep Hygiene Information | Total
Number analyzed (Participants) | 48 | 36 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] — Years
  years | 58.5 (12.7) | 58.7 (14.7) | 58.6 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 39
  Male | 31 | 14 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 48 | 36 | 84
Time since most recent stroke, years [Mean (Standard Deviation); unit: years] | 6 (5) | 6 (5) | 6 (5)

OUTCOME MEASURES:

1. Primary Outcome: Sleep Condition Indicator Score at Post-intervention, Adjusted for Baseline Score and Sex
Description: Self-reported sleep quality questionnaire, range 0-32, higher numbers indicate better sleep quality Assessed at baseline and post-intervention. Outcome is post-intervention score after adjustment for baseline score and sex using Analysis of Covariance
Time Frame: 8 weeks
Population: Intention to treat population, using multiple imputation. Mean and standard deviation are pooled across original (complete case) data and 5 imputations
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Digital CBT-I | Sleep Hygiene Information
Number analyzed (Participants) | 48 | 36
score on a scale | 18.06 [16.47 to 19.66] | 14.72 [13.05 to 16.39]
Statistical Analysis 1: Comparison: Digital CBT-I vs Sleep Hygiene Information; Test type: Superiority; p < 0.021, ANCOVA — p values are calculated for original data (complete case) and each of the 5 imputed datasets. The p value range was 0.002 - 0.020. This is not multiple statistical analyses- it is just one with multiple imputations; Degrees of freedom for original data (complete case): 1,64. Degrees of freedom for imputed datasets: 1,80; Mean Difference (Final Values) = 3.35

2. Secondary Outcome: Sleep Condition Indicator Score at 8 Week Follow up Adjusted for Baseline Score
Description: Self-reported sleep quality questionnaire, range 0-32, higher scores indicate better sleep quality. Assessed at baseline and 8 week follow up. Outcome is follow up score after adjustment for baseline score using Analysis of Covariance.
Time Frame: 16 weeks
Population: Complete case analysis
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Digital CBT-I | Sleep Hygiene Information
Number analyzed (Participants) | 34 | 33
score on a scale | 18.9 [16.8 to 21.0] | 16.0 [13.9 to 18.2]
Statistical Analysis 1: Comparison: Digital CBT-I vs Sleep Hygiene Information; Test type: Superiority; p = 0.059, ANCOVA; ANCOVA of score at 8 week follow up with baseline score as covariate, effect of group; Mean Difference (Final Values) = 2.86, 95% CI 2-sided [-.106 to 5.822]

3. Secondary Outcome: Sleep Fragmentation, Assessed at Post-intervention Adjusted for Baseline
Description: Sleep fragmentation assessed using actigraphy. Higher values indicate more disrupted (worse) sleep. The minimum value is 0. There is no specified maximum value. According to the manual for the software which does the calculation the definition of sleep fragmentation index is "the sum of the Mobile time (%)' and the 'Immobile bouts <=1min (%)".There are no units associated with sleep fragmentation. The values are never presented in the literature or elsewhere as a percentage and therefore they are not presented as a percentage here. Assessed at baseline and post-intervention. Outcome is post-intervention score after adjustment for baseline score using Analysis of Covariance.
Time Frame: 8 weeks
Population: Complete case analysis population
Measure: Mean (95% Confidence Interval); unit: index (no units)
Arm/Group | Digital CBT-I | Sleep Hygiene Information
Number analyzed (Participants) | 32 | 27
index (no units) | 30.8 [27.6 to 34.1] | 32.1 [28.6 to 35.6]
Statistical Analysis 1: Comparison: Digital CBT-I; Test type: Superiority; p = 0.596, ANCOVA; ANCOVA of sleep fragmentation at post-intervention with baseline as covariate, effect of group; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-3.5 to 6.0]

4. Secondary Outcome: Sleep Fragmentation at 8 Week Follow up Adjusted for Baseline
Description: Sleep fragmentation assessed using actigraphy. Higher values indicate more disrupted (worse) sleep. The minimum value is 0. There is no specified maximum value. According to the manual for the software that does the calculation, the definition of sleep fragmentation index is "the sum of the Mobile time (%)' and the 'Immobile bouts <=1min (%)".There are no units associated with sleep fragmentation. The values are never presented in the literature or elsewhere as a percentage and therefore they are not presented as a percentage here. Assessed at baseline and 8 week follow up. Outcome is follow up score after adjustment for baseline score using Analysis of Covariance
Time Frame: 16 weeks
Population: Complete case analysis population
Measure: Mean (95% Confidence Interval); unit: index (no units)
Arm/Group | Digital CBT-I | Sleep Hygiene Information
Number analyzed (Participants) | 32 | 27
index (no units) | 29.3 [26.5 to 32.0] | 33.8 [30.8 to 36.8]
Statistical Analysis 1: Comparison: Digital CBT-I vs Sleep Hygiene Information; Test type: Superiority; p = 0.031, ANCOVA; ANCOVA of sleep fragmentation at 8 week follow up with baseline as covariate, effect of group; Mean Difference (Final Values) = 4.5, 95% CI 2-sided [.431 to 8.612]

5. Secondary Outcome: Wake After Sleep Onset at Post-intervention Adjusted for Baseline
Description: Wake after sleep onset assessed using actigraphy, higher values (minutes) indicate more disrupted sleep. Assessed at baseline and post-intervention. Outcome is post-intervention score after adjustment for baseline score using Analysis of Covariance
Time Frame: 8 weeks
Population: Complete case analysis population
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Digital CBT-I | Sleep Hygiene Information
Number analyzed (Participants) | 32 | 27
minutes | 53 [47 to 59] | 54 [48 to 60]
Statistical Analysis 1: Comparison: Digital CBT-I vs Sleep Hygiene Information; Test type: Superiority; p = 0.885, ANCOVA; ANCOVA of wake after sleep onset post-intervention with baseline as covariate, effect of group; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-7.8 to 9.1]

6. Secondary Outcome: Wake After Sleep Onset at 8 Week Follow up Adjusted for Baseline
Description: Wake after sleep onset assessed using actigraphy, higher values (minutes) indicate more disrupted sleep. Assessed at baseline and 8 week follow up. Outcome is follow up score after adjustment for baseline score using Analysis of Covariance.
Time Frame: 16 weeks
Population: complete case analysis population
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Digital CBT-I | Sleep Hygiene Information
Number analyzed (Participants) | 32 | 27
minutes | 49 [43 to 55] | 57 [50 to 63]
Statistical Analysis 1: Comparison: Digital CBT-I vs Sleep Hygiene Information; Test type: Superiority; p = 0.077, ANCOVA; ANCOVA of wake after sleep onset at 8 week follow up with baseline as covariate, effect of group; Mean Difference (Final Values) = 8, 95% CI 2-sided [-1 to 17]

7. Secondary Outcome: Change in Sleep Onset Latency
Description: Sleep onset latency assessed using online sleep diary, higher values indicate poorer sleep quality
Time Frame: 8 weeks
Population: complete case analysis population
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Digital CBT-I | Sleep Hygiene Information
Number analyzed (Participants) | 34 | 32
minutes | 18 [13 to 24] | 28 [23 to 34]
Statistical Analysis 1: Comparison: Digital CBT-I vs Sleep Hygiene Information; Test type: Superiority; p = 0.014, ANCOVA; ANCOVA of sleep onset latency (median of 7 nights) at end of intervention with baseline as covariate, effect of group; Mean Difference (Final Values) = 10, 95% CI 2-sided [2 to 18]

8. Secondary Outcome: Self-reported Depression Post-intervention, Assessed as PHQ9 Score at Post-intervention Adjusted for Baseline
Description: PHQ9 score, range 0-20, higher values indicate more depressive symptoms. Assessed at baseline and post-intervention. Outcome is post-intervention score after adjustment for baseline score using Analysis of Covariance
Time Frame: 8 weeks
Population: complete case analysis population
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Digital CBT-I | Sleep Hygiene Information
Number analyzed (Participants) | 35 | 33
score on a scale | 5.9 [4.7 to 7.1] | 7.7 [6.6 to 8.9]
Statistical Analysis 1: Comparison: Digital CBT-I vs Sleep Hygiene Information; Test type: Superiority; p = 0.03, ANCOVA; ANCOVA of PHQ9 score post-intervention with baseline as covariate, effect of group; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [.18 to 3.5]

9. Secondary Outcome: Self-reported Depression at 8 Week Follow up, Assessed as PHQ9 Score at 8 Week Follow up Adjusted for Baseline
Description: PHQ9 score, range 0-20, higher values indicate more depressive symptoms. Assessed at baseline and 8 week follow up. Outcome is follow up score after adjustment for baseline score using Analysis of Covariance
Time Frame: 16 weeks
Population: complete case analysis population
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Digital CBT-I | Sleep Hygiene Information
Number analyzed (Participants) | 34 | 33
score on a scale | 5.93 [4.43 to 7.43] | 8.22 [6.7 to 9.75]
Statistical Analysis 1: Comparison: Digital CBT-I vs Sleep Hygiene Information; Test type: Superiority; p = 0.036, ANCOVA; ANCOVA of PHQ9 score at 8 week follow up with baseline as covariate, effect of group; Mean Difference (Final Values) = 2.29, 95% CI 2-sided [.149 to 4.44]

10. Secondary Outcome: Self-reported Anxiety at Post-intervention, Assessed as GAD7 Score Post-intervention Adjusted for Baseline
Description: GAD7 score, range 0-21, higher values indicate more anxiety symptoms. Assessed at baseline and post-intervention. Outcome is post-intervention score after adjustment for baseline score using Analysis of Covariance
Time Frame: 8 weeks
Population: complete case analysis population
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Digital CBT-I | Sleep Hygiene Information
Number analyzed (Participants) | 35 | 33
score on a scale | 5.28 [4.14 to 6.42] | 6.90 [5.72 to 8.06]
Statistical Analysis 1: Comparison: Digital CBT-I vs Sleep Hygiene Information; Test type: Superiority; p = 0.054, ANCOVA; ANCOVA of GAD7 post-intervention, with baseline as covariate, effect of group; Mean Difference (Final Values) = 1.61, 95% CI 2-sided [-0.03 to 3.25]

11. Secondary Outcome: Self-reported Anxiety at 8 Week Follow up, Assessed as GAD7 Score at 8 Week Follow up Adjusted for Baseline
Description: GAD7 score, range 0-21, higher values indicate more anxiety symptoms. Assessed at baseline and 8 week follow up. Outcome is follow up score after adjustment for baseline score using Analysis of Covariance
Time Frame: 16 weeks
Population: complete case analysis population
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Digital CBT-I | Sleep Hygiene Information
Number analyzed (Participants) | 34 | 33
score on a scale | 5.66 [4.41 to 6.91] | 6.75 [5.48 to 8.01]
Statistical Analysis 1: Comparison: Digital CBT-I vs Sleep Hygiene Information; Test type: Superiority; p = 0.229, ANCOVA; ANCOVA of GAD7 at 8 week follow up, with baseline as covariate, effect of group; Mean Difference (Final Values) = 1.09, 95% CI 2-sided [-.70 to 2.87]

12. Secondary Outcome: Stroke Specific Quality of Life, Assessed as SIS Index Post-intervention Adjusted for Baseline
Description: SIS-8 index, range 0-100, higher values less impact of stroke on quality of life. Assessed at baseline and post-interventin. Outcome is post-intervention score after adjustment for baseline score using Analysis of Covariance
Time Frame: 8 weeks
Population: complete case analysis population
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Digital CBT-I | Sleep Hygiene Information
Number analyzed (Participants) | 35 | 33
score on a scale | 51.8 [49.0 to 54.6] | 50.4 [47.5 to 53.3]
Statistical Analysis 1: Comparison: Digital CBT-I vs Sleep Hygiene Information; Test type: Superiority; p = 0.502, ANCOVA; ANCOVA of SIS index at post-intervention, with baseline as covariate, effect of group; Mean Difference (Final Values) = -1.39, 95% CI 2-sided [-5.51 to 2.73]

13. Secondary Outcome: Stroke Specific Quality of Life at 8 Week Follow up, Assessed as SIS Index at 8 Week Follow up Adjusted for Baseline
Description: SIS-8 index, range 0-100, higher values indicate less impact of stroke on quality of life. Assessed at baseline and 8 week follow up. Outcome is follow up score after adjustment for baseline score using Analysis of Covariance
Time Frame: 16 weeks
Population: complete case analysis population
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Digital CBT-I | Sleep Hygiene Information
Number analyzed (Participants) | 34 | 33
score on a scale | 52.0 [49.3 to 55.0] | 52.1 [49.5 to 54.8]
Statistical Analysis 1: Comparison: Digital CBT-I vs Sleep Hygiene Information; Test type: Superiority; p = 0.924, ANCOVA; ANCOVA of SIS index at 8 week follow up, with baseline as covariate, effect of group; Mean Difference (Final Values) = .183, 95% CI 2-sided [-3.63 to 4.0]

14. Other Pre Specified Outcome: Cost Effectiveness
Description: Assessed as incremental cost effectiveness ratio, using EQ-5D-5L, range 0-5 for each dimension, higher values indicate more problems
Time Frame: 16 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events could be reported to the research team at any time during the intervention or over the 8 weeks following the intervention. The length of the intervention was not prescribed, but on average it lasted 77 days. Therefore on average adverse events could be reported over a 19 week timescale, being 11 weeks (77 days average) for the intervention period plus the 8 week follow up period.
Arm/Group | Digital CBT-I | Sleep Hygiene Information
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT04272892/Prot_SAP_ICF_000.pdf